CLINICAL TRIAL: NCT04342767
Title: The Effectiveness of a Mechanical Debridement Instrument in Reducing Bioburden in Chronic Wounds
Status: Completed | Type: Observational
Sponsor: SerenaGroup, Inc. (Network)
Collaborators: MDM Wound Ventures, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: EZ-1
Record Dates: First submitted 2020-04-07; First posted 2020-04-13 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Acute Wounds; Chronic Wounds

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: EZ Debride® — EZ Debride ® is intended for the mechanical debridement of topical wounds including partial and full thickness wounds, pressure ulcers, venous ulcers, diabetic ulcers, chronic vascular ulcers, surgical wounds (donor sites/grafts, post Mohs' surgery, post-laser surgery, podiatric, wound dehiscence) trauma wounds (abrasions, lacerations, second-degree burns and skin tears), draining wounds and tunnelled /undermined wounds.

SUMMARY:
This prospective clinical trial will compare the bacterial burden in the wound bed and on the periwound skin before and after mechanical debridement with EZ Debride using fluorescence imaging.

After consenting, the ulcers of eligible subjects are measured, photographed and undergo the MolecuLight imaging procedure (MLiX). The ulcer is mechanically debridement with the EZ Debride device after which a second MLiX procedure is performed. The investigator will then compare the two images.

DETAILED DESCRIPTION:
Acute and chronic wounds burden healthcare systems across the globe. In the United States the cost of nonhealing wounds approximates 100 billion dollars.1-3 The presence of bacteria in and around the wound impedes wound healing. Clinicians treat elevated wound bacterial levels with mechanical and sharp debridement, topical antiseptics and systemic antibiotics. However, evidence on the best methods to reduce bacterial load is lacking. The EZ-1 clinical trial will utilize the latest fluorescence imaging technology to investigate whether mechanical debridement using the EZ Debride® tool reduces bacterial burden.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with acute or chronic wounds that have been present for a minimum of 4 weeks.
2. A signed and dated informed consent form.
3. Subject is willing and able to comply with instructions and scheduled visits.

Exclusion Criteria:

1. The Subject has other concurrent conditions that in the opinion of the Investigator may compromise subject safety.
2. The subject's wound has not been present for at least 4 weeks.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute or chronic wounds
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Change in Bacterial Bioburden | Before and After Mechanical debridement within 1 hour
  The reduction in bacterial bioburden following mechanical wound debridement as determined by the MolecuLight Procedure (MLiX).

SECONDARY OUTCOMES:
Pain Score | Before, during, and after mechanical debridement within 1 hour
  Pain scores (PEG) before, during and after mechanical debridement. Pain intensity of the reference ulcer is assessed before and after any wound cleansing using the PEG score
  PEG Scale Assessing Pain Intensity and Interference (Pain, Enjoyment, General Activity). The PEG scale is a validated pain scoring system. It consists of three 1-10 rating scales: numerical, enjoyment of life and general activity. The subject indicates a numerical value that best represents the pain intensity at ulcer site on a scale of 0 to 10 anchored by word descriptors at each end, as "no pain" on the left side and "Pain as bad as you can imagine" on the right side of the number line. The number 0 represents "no pain", the number 5 represents "moderate pain" and the number 10 represents the "worst possible pain".
Adverse Events | During debridement
  Adverse events associated with mechanical debridement.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Serena, MD,FACS, Principal Investigator — SerenaGroup, Inc.
Locations (1):
- Serena Group Research Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No